CLINICAL TRIAL: NCT07384377
Title: A Phase III Trial to Evaluate the Efficacy and Safety of JSKN003 Versus Physician Choiced Treatment in Patients With HER2-positive and Advanced Colorectal Cancer Who Had Failed to Respond to Oxaliplatin, 5-Fu, and Irinotecan
Brief Title: JSKN003 Versus Physician Choiced Treatment in Patients With HER2-positive and Advanced Colorectal Cancer Who Had Failed to Respond to Oxaliplatin, 5-Fu, and Irinotecan
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-005
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Colorectal Cancer
MeSH Terms: interventions — regorafenib; HMPL-013

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, multi-center Phase III clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JSKN003 (Active Comparator)
  Interventions: Drug: JSKN003
- Physician choiced treatment (Active Comparator)
  Interventions: Drug: Physician choiced treatment, include: TAS-102, Regorafenib, Fruquintinib.

INTERVENTIONS:
Drug: JSKN003 — JSKN003 (6.3 mg/kg) was administered intravenously on the first day of each cycle, once every 3 weeks (Q3W).
  Arms: JSKN003
Drug: Physician choiced treatment, include: TAS-102, Regorafenib, Fruquintinib. — TAS-102(35 mg/m2, maximum 80 mg per dose), twice daily (BID), once every 4 weeks (Q4W); or Regorafenib 160mg, once daily (QD), once every 4 weeks (Q4W); or Fruquintinib 5mg once daily (QD), once every 4 weeks (Q4W).
  Arms: Physician choiced treatment

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of JSKN003 Versus Physician Choiced Treatment in Patients With HER2-positive and Advanced Colorectal Cancer Who had Failed to Respond to Oxaliplatin, 5-Fu, and Irinotecan subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old.
* Unresectable locally advanced or distant metastatic BRAFV600E wild-type colorectal cancer diagnosed histologically or cytologically.
* After treatment with oxaliplatin, 5-fluorouracil (such as 5-FU, Capecitabine) , irinotecan (DMMR/MSI-H subjects also need anti-PD-1/PD-L1 antibody treatment failure).
* HER2-positive (defined as IHC3+ or IHC 2+/FISH +).
* According to the response evaluation criteria for solid tumors (RECIST 1.1), having at least one assessable lesion, assessable lesions should not have received local treatment such as radiotherapy (lesions located within the previously treated area may also be targeted if progression is confirmed).
* ECOG PS of 0-1.
* Expected survival ≥ 3 months.
* Participants with adequate organ functions.
* Female and male patients of childbearing age agree to take adequate contraceptive measures during and upon completion of the study for 7 months after the last dose. Female participants of childbearing age must have a negative blood pregnancy test within 7 days before the first dose or randomization.
* Voluntarily agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Participants who have previously been treated with an anti-HER2 ADC loaded with topoisomerase I inhibitors.
* Participants with brain metastasis or spinal cord compression at screening.
* Previous antineoplastic therapy toxicities did not revert to a CTCAE v5.0 grade rating of ≤1.
* There are obvious clinical manifestations of gastrointestinal abnormalities, including but not limited to: having experienced intestinal obstruction or symptoms and signs of intestinal obstruction within 3 months prior to administration; having had gastrointestinal perforation, gastrointestinal fistula, or intra-abdominal abscess within 3 months prior to administration; having experienced gastrointestinal bleeding of CTCAE grade ≥ 3 within 3 months prior to administration, or having had gastrointestinal bleeding within the previous 1 month.
* Participants who have undergone major surgery or had invasive intervention within 28 days before the randomization. Or those who plan to undergo systematic or local tumor resection during the trial.
* Participate in another clinical trial, unless it is an observational (non-intervention) clinical trial or is in the follow-up period of an intervention trial.
* Participants who have used any Chinese herbal medicine or Chinese patent medicine approved by the national drug regulatory authority for its anti-cancer properties within the previous 14 days (regardless of the type of cancer); have received palliative radiotherapy within the 14 days prior to randomization; have received systemic anti-tumor treatment within 4 weeks or 5 half-life (whichever is shorter but at least 2 weeks) prior to randomization.
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
* Participants who have active bacterial, fungal or viral infections 14 days before the randomization.
* Within the 14 days before the randomization, participants who had a situation where there was an uncontrollable need for frequent drainage or medical intervention in the serous cavity effusion.
* Participant with positive hepatitis B surface antigen (HBsAg) and HBV-DNA is higher than 500 IU/mL (or 2500 copies/ml) (whichever is lower) ; Participants with positive for hepatitis C (HCV) antibody and HCV-RNA is higher than 1000 copies/ml or UNL (whichever is lower).
* Has activity or a history of interstitial lung disease at any stage and/or pulmonary function injury, a history of interstitial pneumonia requiring hormone therapy, or the imaging cannot rule out suspected interstitial lung disease/pneumonia at screening.
* Has a history of severe cardiovascular disease.
* History of any other malignant tumors within 5 years.
* Pregnant or breastfeeding women.
* Otherwise considered inappropriate for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Progressive Free Survive (PFS) assessed by Independent Review Committee | Every 6 weeks, up to 3 years

SECONDARY OUTCOMES:
Progressive Free Survive (PFS) assessed by the Investigator | Every 6 weeks, up to 3 years
Objective response rate (ORR) assessed by the Investigator or IRC | Every 6 weeks, up to 3 years
Duration of Response (DOR) assessed by the Investigator or IRC | Every 6 weeks, up to 3 years
Overall Survival (OS) | Up to approximately 3 years
Incidence and severity of TEAE and SAE | Up to approximately 3 years
Blood concentration of JSKN003 | Up to approximately 3 years
Blood concentration of total antibodies for JSKN003 | Up to approximately 3 years
Blood concentration of free toxins for JSKN003 | Up to approximately 3 years
Anti-drug antibodies (ADA) related to JSKN003 | Up to approximately 3 years